CLINICAL TRIAL: NCT00935389
Title: Prospective Control Study of TW in the Treatment of LN Type V With Gross Proteinuria
Brief Title: Prospective Study of TW in the Treatment of LN Type V With Gross Proteinuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Nanjing University School of Medicine, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0903
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2009-07

CONDITIONS: Lupus Nephritis; Proteinuria; CTX
MeSH Terms: conditions — Lupus Nephritis; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- immunosuppressor (Experimental): TW 30mg,q.d.*3 months and reduced into 20mg b.i.d
  Interventions: Drug: tripterygium glycosides

INTERVENTIONS:
Drug: tripterygium glycosides — The onset dosage should be 30mg/q.d. and can be reduced into 20mg b.i.d if CR obtained in 3 months. Without CR in 3 months, the dosage of 90mg/d will last for another 3 months and then reduced to 60mg/d.
  Other Names: TW

SUMMARY:
The purpose of this study is to analyze the clinical effects and adverse reactions of tripterygium glycosides (TW) and CTX in LN-V patients with gross proteinuria.

DETAILED DESCRIPTION:
Compared with cyclophosphamide(CTX), to analyze the clinical effects and adverse reactions of tripterygium glycosides (TW) in LN-V patients with gross proteinuria.

ELIGIBILITY:
Inclusion Criteria:

1. SLE patients aging 18-60 years, all of whom comply to the ISN/RPS classification.
2. Urine protein≥3.0g/24h, Alb<30g/L and Scr<1.5mg/dL.
3. All cases are type IV, confirmed by renal biopsy.
4. All patients sign the informed consent and be willing to follow-up on time

Exclusion Criteria:

1. Accepted drug therapy, such as CTX MMF CsA FK506 or TW more than 2 weeks in the latest 3 months.
2. Scr level above 1.5mg/dL, lasts more than 3 months.
3. Heart, lung or central nervous systems involved or combined with severe infection.
4. With liver function abnormal, ALT or AST being two times above the normal.
5. Pregnant women or patients still in lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To analyze the clinical effects of tripterygium glycosides (TW) in LN-V patients with gross proteinuria. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Hu Weixin, Doctor, Principal Investigator — Jinling Hospital, China
Locations (2):
- China (2):
  - Research Institute of Nephrology, Jinling Hospital, Nanjing, Jiangsu
  - Research Institute of Nephrology,Jinling Hospital, Nanjing, Jiangsu